CLINICAL TRIAL: NCT00728520
Title: A Phase II Trial With Azacitidine Single Agent in Newly Diagnosed Acute Myelogenous Leukemia (AML) Veterans Administration (VA) Elderly Patients Who Are Ineligible for Standard Induction Therapy: A Department of Veterans Affairs Multi-Site Study
Brief Title: Trial With Azacitidine in Newly Diagnosed Acute Myelogenous Leukemia (AML) Veterans Administration (VA) Elderly Patients Not Eligible for Standard Induction Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Suman Kambhampati, MD, Kansas City Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SK0010
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Acute Myeloid Leukemia; Elderly
Keywords: Leukemia; Azacitidine; Untreated; Elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 75 mg/m2 daily IV or subcutaneously (SQ) for 5 days, every 4 weeks for a minimum of 4 cycles.
  Other Names: Vidaza

SUMMARY:
The drug that will be used in this study is called Azacitidine. Azacitidine belongs to a group of drugs which may restore normal control in cancer cells by affecting the genes and proteins in the body. Azacitidine is approved by the FDA for the treatment of Myelodysplastic Syndrome (MDS), a pre-leukemic bone marrow disease. The purpose of this study is to find out what effect the drug Azacitidine has on Acute Myeloid Leukemia (AML) in elderly patients.

DETAILED DESCRIPTION:
Prior to starting treatment individuals being considered for this study will be evaluated to determine if they are eligible to participate in the study. There are certain prestudy test that are required: physical exam, blood tests, ECG, chest x-ray, bone marrow aspirate and biopsy to confirm the diagnosis of AML.

Treatment regimen consists of Azacitidine IV/SQ on days 1-5 every 28 days. If the Azacitidine is given IV it will be given over 15-40 minutes. The treatment will be given for a minimum of 4 treatment cycles. Blood samples will be taken every week to monitor for side effects of the Azacitidine. A bone marrow aspirate will be done every 3-4 months to determine the response to the study drug or until the disease progresses. There is also a quality of life questionnaire that will be completed at the beginning of the study and every 4 weeks while on the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML
* Elderly patients with denovo AML or secondary AML evolving from MDS in patient >/= 60 who decline chemotherapy or those who are not currently candidates for induction chemotherapy
* Stable WBC <10 x 109 and not requiring hydroxyurea, chemotherapy or leukapheresis for >4 weeks
* No corticosteroids, hydroxyurea, low-dose cytarabine, interferon, ir retinoids within 1 month
* No prior decitabine
* No valproic acid or other histone deacetylase inhibitor for at least 2 weeks
* No G-CSF, or GM-CSF or Erythropoetin within 1 month of study entry
* No investigational agents within 28 days
* ECOG performance status </= 2 or KPS >/= 60%
* Life expectancy > 2 months
* Normal organ function = Total bilirubin </= 1.5 x ULN, AST/ALT </= 2.5 x ULN
* Creatinine within normal limits or creatinine clearance >/= 60ml/min
* Signed informed consent

Exclusion Criteria:

* Patients with t(15;17) or M3-AML
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to study entry, or who have not recovered from adverse effects of agents administered earlier
* Patients with CNS involvement of AML
* History of allergic reactions attributed to Azacitidine or compounds of similar chemical used in this study
* Pregnancy
* Other serious medical or psychiatric illness which would limit survival to < 3 months or prevent the granting of informed consent or lead to situations that would limit compliance with study requirements
* Known positive serology for HIV, HIV positive patients with anti-retroviral therapy are ineligible
* Active systemic bacterial, fungal or viral infection
* Patients with severe complications of the leukemia including but not limited to active infection, uncontrolled infection, pneumonia, hypoxia, and shock
* Patients with advanced hepatic tumors
* Patients with poor history of medical compliance
* Patients with known platelet refractoriness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
overall response rates, duration of response, toxicities | Starting 4 weeks after treatment, during the entire study duration, and upon study completion

SECONDARY OUTCOMES:
leukemia free survival, overall survival, quality of life, assess biomarkers and predictive markers for Azacitidine responsiveness in elderly AML patients | During the entire duration of the study and after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Amit Verma, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Kansas City Veterans Affairs Medical Center, Kansas City, Missouri, United States